CLINICAL TRIAL: NCT01301274
Title: Randomized, Controlled, Double Blinded, Clinical Trial: 0.9% NaCl/Dextrose 5% vs 0.45% NaCl/Dextrose 5% as Maintenance Intravenous Fluids in Critically Ill Children
Brief Title: 0.9% NaCl/Dextrose 5% vs 0.45% NaCl/Dextrose 5% as Maintenance Intravenous Fluids in Critically Ill Children
Acronym: NaCrICh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HGNPE-20-2011
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Results first posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Hyponatremia
Keywords: hyponatremia; maintenance solutions; pediatrics
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypotonic (Active Comparator): Subjects in this arm will receive 0.45% NaCl/5% dextrose intravenous maintenance fluids.
  Interventions: Drug: hypotonic
- Isotonic (Experimental): Subjects in this arm will receive 0.9% NaCl/5% dextrose intravenous maintenance fluids.
  Interventions: Drug: isotonic

INTERVENTIONS:
Drug: hypotonic — 0.45% NaCl/5% dextrose IV maintenance fluids
  Other Names: half saline/5% dextrose
  Arms: Hypotonic
Drug: isotonic — 0.9% NaCl/5% dextrose IV maintenance fluids
  Other Names: normal saline/5% dextrose
  Arms: Isotonic

SUMMARY:
The primary objective of this study is to compare the mean serum sodium after 48 hours of therapy with either 0.45% NaCl/dextrose 5% or 0.9% NaCl/dextrose 5%, in critically ill children requiring IV maintenance fluid administration.

DETAILED DESCRIPTION:
In patients without possibilities of oral intake, maintenance fluids provide electrolytes and water. Since the original descriptions by Holliday and Segar, the recommended standard maintenance solutions are based on "physiological needs", containing 30-50 mEq/L of sodium.

However hyponatremia has become increasingly recognized in hospitalized children suggesting that Holliday and Segar's recommendations are frequently inappropriately applied.

It has been described augmented intersticial lung water in patients receiving hypotonic maintenance solutions. Also, hyponatremia has been demonstrated in post-surgery critically ill children receiving hypotonic maintenance solutions.

More over, non-physiologic antidiuretic hormone (ADH) secretion has been described in the great majority of hospitalized children due to nausea, stress, pain, and/or surgical interventions.

It has been suggested that isotonic 0.9% NaCl/dextrose 5% should be the standard maintenance intravenous (IV) solution, to avoid the development of hyponatremia.

There are not studies in critically ill children evaluating the effect of isotonic solutions on sodium levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 month to 18 years
* ICU stay >24 hours
* Normal seric sodium (135 - 145 mEq/L).
* Requirement of IV maintenance solutions >80% total fluids intake

Exclusion Criteria:

* Patients with diagnoses of renal failure (serum creatinine >1 g/dl in <3 years old children, >1,5 in >3 years), hepatic failure with ascitis and portal hypertension, adrenal failure, nephrotic - nephritic syndrome, Kawasaki disease, sickle cell anemia, Syndrome of inappropriate antidiuretic hormone secretion, diabetes insipidus,metabolic disease.
* Diuretics use in the first 48 hours thereafter indicated IV solutions.
* Plasma glucose is >200 mg%.
* Any patients requiring IV fluids therapy different that maintenance (total parenteral nutrition, hyperhydration).

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Facundo A Jorro, MD, Principal Investigator — Hospital General de Niños Pedro de Elizalde; Gustavo De Baisi, MD, Study Director — Hospital General de Niños Pedro de Elizalde; Susana Bengoa, Principal Investigator — Hospital General de Niños Pedro de Elizalde
Locations (1):
- Hospital General de Niños Pedro de Elizalde, Buenos Aires, Argentina

REFERENCES:
- [Background] HOLLIDAY MA, SEGAR WE, LUKENBILL A, VALENCIA RM, DURELL AM. Variations in muscle electrolyte composition due to sampling and to aging. Proc Soc Exp Biol Med. 1957 Aug-Sep;95(4):786-8. doi: 10.3181/00379727-95-23364. No abstract available. PMID 13465804
- [Background] Burrows FA, Shutack JG, Crone RK. Inappropriate secretion of antidiuretic hormone in a postsurgical pediatric population. Crit Care Med. 1983 Jul;11(7):527-31. doi: 10.1097/00003246-198307000-00009. PMID 6861500
- [Background] Eulmesekian PG, Perez A, Minces PG, Bohn D. Hospital-acquired hyponatremia in postoperative pediatric patients: prospective observational study. Pediatr Crit Care Med. 2010 Jul;11(4):479-83. doi: 10.1097/PCC.0b013e3181ce7154. PMID 20124948
- [Background] Choong K, Kho ME, Menon K, Bohn D. Hypotonic versus isotonic saline in hospitalised children: a systematic review. Arch Dis Child. 2006 Oct;91(10):828-35. doi: 10.1136/adc.2005.088690. Epub 2006 Jun 5. PMID 16754657
- [Derived] Jorro Baron FA, Meregalli CN, Rombola VA, Bolasell C, Pigliapoco VE, Bartoletti SE, Debaisi GE. Hypotonic versus isotonic maintenance fluids in critically ill pediatric patients: a randomized controlled trial. Arch Argent Pediatr. 2013 Jul-Aug;111(4):281-7. doi: 10.5546/aap.2013.eng.281. English, Spanish. PMID 23912284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Intensive Care Unit without cardiovascular patients, since 01/02/2011 until 01/11/2011
Pre-assignment Details: 251 admitted patients to ICU, 97 eligible patients, 9 patients did not give consent, 22 were not randomized by treatment physician
Period: Overall Study
Arm/Group | Hypotonic | Isotonic
Started | 34 | 32
Completed | 32 | 31
Not Completed | 2 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypotonic | Isotonic | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 32 | 66
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 3 (4.7) | 1.2 (3.2) | 2.2 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  Argentina | 34 | 32 | 66

OUTCOME MEASURES:

1. Primary Outcome: Serum Sodium Levels in Both Groups
Description: Mean serum sodium level of each group will be compared at baseline and in the first 48 hours of IV fluid infusion
Time Frame: first 48 hours
Measure: Mean (Standard Deviation); unit: mEq/L
Groups:
- Hypotonic Arm: patients who received for maintenance solution 0.45% ClNa in Dx 5%
- Isotonic Arm: Patients who received for maintenance solution 0.9% ClNa in Dx 5%
Arm/Group | Hypotonic Arm | Isotonic Arm
Number analyzed (Participants) | 32 | 31
mEq/L | 137.8 (4.3) | 140.0 (4.1)
Statistical Analysis 1: Comparison: Hypotonic Arm vs Isotonic Arm; Test type: Non-Inferiority or Equivalence — beta error 20%, alfa error 5%, diminished 2 mEq/L between groups; p = 0.04, t-test, 2 sided

2. Secondary Outcome: Mortality at 28 Days
Description: Mortality in both groups will be compared 28 days after admission
Time Frame: 28 days after admission
Population: The analysis was per intention to treat
Measure: Number; unit: participants
Groups:
- Hypotonic Arm: patients who received maintenance solution 0.45% ClNa in Dx 5%
- Isotonic Arm: patients who received maintenance solution 0.9% ClNa in Dx 5%
Arm/Group | Hypotonic Arm | Isotonic Arm
Number analyzed (Participants) | 32 | 31
participants | 3 | 0
Statistical Analysis 1: Comparison: Hypotonic Arm vs Isotonic Arm; Test type: Superiority or Other; p = 0.081, Chi-squared — without adjust

3. Secondary Outcome: Mechanical Ventilation Free Days at 28 Day of Admission
Description: mechanical ventilation free days at the first 28 day of starting mechanical ventilation, if the patient died the corresponding value is zero.
Time Frame: first 28 day after starting mechanical ventilation
Measure: Mean (Standard Deviation); unit: days
Groups:
- Hypotonic Arm: patients who received fro maintenance solution ClNa 0.45% in Dx 5%
- Isotonic Arm: patients who received for maintenance solution ClNa 0.9% in Dx 5%
Arm/Group | Hypotonic Arm | Isotonic Arm
Number analyzed (Participants) | 32 | 31
days | 19.9 (7.9) | 21.5 (6.6)
Statistical Analysis 1: Comparison: Hypotonic Arm vs Isotonic Arm; Test type: Superiority or Other; p = 0.396, t-test, 2 sided

4. Secondary Outcome: ICU Length of Stay
Description: ICU length of stay (in days)
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: days
Groups:
- Hypotonic Arm; Isotonic Arm: patients who received for maintenance solution ClNa 0.9% in Dx 5%
Arm/Group | Hypotonic Arm | Isotonic Arm
Number analyzed (Participants) | 32 | 31
days | 8.5 (5.5) | 11.9 (11.5)
Statistical Analysis 1: Comparison: Hypotonic Arm vs Isotonic Arm; Test type: Superiority or Other; p = 0.129, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: until they were receiving the maintenance solution, mean time 24 hours up to 48 hours. The adverse events were collected up to PICU discharged, mean time 7.4 days, except mortality up to 28 days.
Arm/Group | Hypotonic | Isotonic
Serious Adverse Events (participants affected / at risk) | 4/34 | 0/32
Other Adverse Events (participants affected / at risk) | 5/34 | 4/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypotonic (N=34) | Isotonic (N=32)
hyponatremia <130 mEq/l (General disorders) | 1 (1) | 0 (0) — serum sodium <130 mEq/l, without symptoms.
Death (General disorders) | 3 (3) | 0 (0) — patient death that occurred between up to 28 days after randomization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypotonic (N=34) | Isotonic (N=32)
Serum sodium < 135 mEq/l (General disorders) | 5 (5) | 4 (4) — serum sodium between 130 - 134,9 mEq/l, without neurological symptoms.

LIMITATIONS AND CAVEATS:
Limitations: Antidiuretic hormone were not measured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes